CLINICAL TRIAL: NCT00232154
Title: An Open-Label Study Of Azithromycin Pharmacokinetics In Sinus Mucosal Tissue And Plasma In Subjects With Chronic Rhinosinusitis Following A Single 2g Dose Of Azithromycin Extended Release For Oral Suspension Or Azithromycin 500mg Tablet Formulation Once Daily For A Maximum Of Three Days
Brief Title: A Study To Measure The Level Of Drug In Nasal Tissue And Blood After Taking A Single 2g Dose Or 500mg Tablets For Up To
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: A0661151
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Azithromycin; Blood Specimen Collection; Hematologic Tests

INTERVENTIONS:
Drug: Zithromax™ (azithromycin) 500mg tablets
Procedure: Endoscopic Sinus Surgery
Procedure: Blood sampling for hematology
Procedure: Blood sampling for plasma chemistry profile
Procedure: Serum pregnancy test (for women of child-bearing potential)

SUMMARY:
To measure the level of drug in nasal tissue and blood after taking a single 2g dose or 500mg tablets for up to 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects considered by the Principal Investigator as an appropriate candidate for endoscopic sinus surgery, e.g., for the removal of the thickened and diseased mucosal tissue that blocks the ostiomeatal complex (OMC).

Exclusion Criteria:

* Known or suspected hypersensitivity or intolerance to any macrolide-like compound, including erythromycin, clarithromycin, azithromycin or telithromycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-11; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of azithromycin in sinus mucosal tissue and plasma in adult subjects after treatment with a single 2 g oral dose of azithromycin extended release for oral suspension or oral azithromycin 500 mg tablet

SECONDARY OUTCOMES:
To assess the safety of azithromycin extended release for oral suspension and azithromycin 500mg tablets.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (14):
  - Pfizer Investigational Site, Alabaster, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Hoover, Alabama
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Elgin, Illinois
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Carrollton, Kentucky
  - Pfizer Investigational Site, La Grange, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661151&StudyName=A+Study+To+Measure+The+Level+Of+Drug+In+Nasal+Tissue+And+Blood+After+Taking+A+Single+2g+Dose+Or+500mg+Tablets+For+Up+To+